CLINICAL TRIAL: NCT02515955
Title: A Randomized, Placebo- and Comparator-controlled, Double-blind, Multiple (Ascending) Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-54175446 in Healthy Male Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-54175446 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107762; 54175446EDI1002 (Other: Janssen-Cilag International NV); 2015-001300-55 (EudraCT Number)
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-54175446
MeSH Terms: interventions — JNJ-54175446; Minocycline; Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 (Experimental): Participants will be receiving either JNJ-54175446 at increasing dose levels using 2 oral formulation as suspension for oral dose once daily from Day 1 to Day 17 or minocycline 100 mg capsule twice daily from Day 1 to Day 17 or placebo matching with JNJ 54175446 once daily from Day 1 to Day 17.
  Interventions: Drug: JNJ-54175446; Drug: Minocycline; Drug: JNJ 54175446 Matching Placebo; Drug: D Amphetamine; Drug: D Amphetamine Matching Placebo
- Cohort 2 (Experimental): Participants will be receiving either JNJ-54175446 at increasing dose levels using 2 oral formulation as suspension for oral dose once daily from Day 1 to Day 17 or minocycline 100 mg capsule twice daily from Day 1 to Day 17 or placebo matching with JNJ 54175446 once daily from Day 1 to Day 17.
  Interventions: Drug: JNJ-54175446; Drug: Minocycline; Drug: JNJ 54175446 Matching Placebo; Drug: D Amphetamine; Drug: D Amphetamine Matching Placebo
- Cohort 3 (Experimental): Participants will be receiving either JNJ-54175446 at increasing dose levels using 2 oral formulation as suspension for oral dose once daily from Day 1 to Day 17 or minocycline 100 mg capsule twice daily from Day 1 to Day 17 or placebo matching with JNJ 54175446 once daily from Day 1 to Day 17.
  Interventions: Drug: JNJ-54175446; Drug: Minocycline; Drug: JNJ 54175446 Matching Placebo; Drug: D Amphetamine; Drug: D Amphetamine Matching Placebo
- Cohort 4 (Experimental): Participants will be receiving either JNJ-54175446 at increasing dose levels using 2 oral formulation as suspension for oral dose once daily from Day 1 to Day 17 or minocycline 100 mg capsule twice daily from Day 1 to Day 17 or placebo matching with JNJ 54175446 once daily from Day 1 to Day 17.
  Interventions: Drug: JNJ-54175446; Drug: Minocycline; Drug: JNJ 54175446 Matching Placebo; Drug: D Amphetamine; Drug: D Amphetamine Matching Placebo
- Cohort 5 (Experimental): Participants will be receiving either JNJ-54175446 at increasing dose levels using 2 oral formulation as suspension for oral dose once daily from Day 1 to Day 17 or minocycline 100 mg capsule twice daily from Day 1 to Day 17 or placebo matching with JNJ 54175446 once daily from Day 1 to Day 17.
  Interventions: Drug: JNJ-54175446; Drug: Minocycline; Drug: JNJ 54175446 Matching Placebo; Drug: D Amphetamine; Drug: D Amphetamine Matching Placebo
- Cohort 6 (Experimental): Participants will be receiving either JNJ-54175446 at increasing dose levels using 2 oral formulation as suspension for oral dose once daily from Day 1 to Day 17 or minocycline 100 mg capsule twice daily from Day 1 to Day 17 or placebo matching with JNJ 54175446 once daily from Day 1 to Day 17.
  Interventions: Drug: JNJ-54175446; Drug: Minocycline; Drug: JNJ 54175446 Matching Placebo; Drug: D Amphetamine; Drug: D Amphetamine Matching Placebo
- Cohort 7 (Experimental): Participants will be receiving either JNJ-54175446 at increasing dose levels using 2 oral formulation as suspension for oral dose once daily from Day 1 to Day 17 or placebo matching with JNJ 54175446 once daily from Day 1 to Day 17.
  Interventions: Drug: JNJ-54175446; Drug: JNJ 54175446 Matching Placebo; Drug: D Amphetamine; Drug: D Amphetamine Matching Placebo
- Cohort 8 (Experimental): Participants will be receiving either JNJ-54175446 at increasing dose levels using 2 oral formulation as suspension for oral dose once daily from Day 1 to Day 17 or placebo matching with JNJ 54175446 once daily from Day 1 to Day 17.
  Interventions: Drug: JNJ-54175446; Drug: JNJ 54175446 Matching Placebo; Drug: D Amphetamine; Drug: D Amphetamine Matching Placebo

INTERVENTIONS:
Drug: JNJ-54175446 — Participants will receive JNJ-54175446, at increasing dose levels using 2 oral formulations i.e. 0.5 mg/ml and 20 mg/ml as suspension for oral dose once daily.
Drug: Minocycline — Participants will receive minocycline 100 mg as capsule twice daily.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6
Drug: JNJ 54175446 Matching Placebo — Participants will receive placebo matching with JNJ 54175446 once daily orally.
Drug: D Amphetamine — Participants will receive 20 mg d-amphetamine (AMPH) 2 hours after administration of study drug (JNJ-54175446/placebo or minocycline/placebo) on Day 7 and Day 10.
Drug: D Amphetamine Matching Placebo — Participants will receive d-amphetamine (AMPH) matching placebo, 2 hours after administration of study drug (JNJ-54175446/placebo or minocycline/placebo) on Day 7 and Day 10.

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacodynamics of JNJ-54175446 after multiple consecutive dose administrations

DETAILED DESCRIPTION:
This will be a randomized, placebo-and comparator-controlled, double-blind, multiple dose study with JNJ-54175446 in healthy male participants. The study will consist of a Screening examination (28 to 6 days prior to dose administration), a baseline 20 mg amphetamine (AMPH) challenge at least 5 days before first dose administration, a double-blind treatment period (18 days; 11 days of dosing with JNJ-54175446, minocycline or placebo; amphetamine (AMPH)/AMPH placebo challenge sequence on Day 7 and Day 10 for each participant), and a follow-up examination between 14 and 21 days after last dose administration. The maximal study duration for each participant will not exceed 9 weeks. Safety, pharmacokinetics (PK) and pharmacodynamics of JNJ-54175446 will be primarily assessed. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI) between 18 and 32 kilogram/meter^2 (kg/m^2), inclusive (BMI = weight/height^2)
* Participants must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) [including QTcF less than or equal to 450 millisecond (ms) (triplicate ECG)] performed at screening and admission to the clinical unit. Minor abnormalities in ECG, which are not considered to be of clinical significance by the investigator, are acceptable. The presence of Left Bundle Branch Block (LBBB), atrioventricular (AV) Block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator [ICD] will lead to exclusion
* Participants must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel [including liver enzymes], hematology, or urinalysis are outside the normal reference ranges, the subject may be included only if the investigator judges the abnormalities to be not clinically significant. This determination must be recorded in the subject's source documents and initialed by the investigator
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug. In addition, their female partner should also use an appropriate method of birth control for at least the same duration

Exclusion Criteria:

* Participant has a history of or current liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances, any inflammatory illness or any other illness that the Investigator considers should exclude the subject
* Participant has a clinically significant (history of) psychiatric illnesses or (history of) psychotic symptoms
* Participant has a family history of relevant psychiatric disorders (first degree) and/or psychotic disorders (first and second degree)
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening
* Participant has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at Screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Baseline up to 14 or 21 days after study drug administration
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Maximum Observed Plasma Concentration (Cmax) | Baseline up to Day 17
  The Cmax is the maximum observed concentration.
Minimum Observed Plasma Concentration (Cmin) | Baseline up to Day 17
  The Cmin is the minimum observed plasma concentration.
Trough Plasma Concentration (Ctrough) | Baseline up to Day 17
  The (Ctrough) is the plasma concentration before dosing or at the end of the dosing interval of any dose other than the first dose in a multiple dosing regimen.
Average Plasma Concentration at Steady State (Cavg,ss) | Baseline up to Day 17
  The Cavg,ss is calculated as area under the plasma concentration-time curve during a dosing Interval (AUC[tau]) divided by the dosing interval (tau).
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Baseline up to Day 17
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Baseline up to Day 17
  The AUCtau is the measure of the plasma drug concentration from time zero to end of dosing interval. It is used to characterize drug absorption.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) | Baseline up to Day 17
  The AUC(0-t) is the area under the plasma concentration-time curve from time zero to any time 't'.
Elimination Half-Life (t1/2) | Baseline up to Day 17
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical trials, Study Director — Janssen-Cilag International NV
Locations (1):
- Leiden, Netherlands